CLINICAL TRIAL: NCT04438018
Title: Towards a Better Understanding of Diabetes Distress, Depression and Poor Glycaemic Control Leading to Personalised Interventions for People With Type 2 Diabetes
Brief Title: Towards a Better Understanding of Diabetes Distress, Depression and Poor Glycaemic Control in T2DM
Acronym: DIA-LINK2
Status: Completed | Type: Observational
Sponsor: Norbert Hermanns (Other)
Collaborators: German Center for Diabetes Research (Other); University of Giessen (Other); Helmholtz Zentrum München (Industry)
Responsible Party: Sponsor-Investigator, Norbert Hermanns, Prof. Dr. phil., Forschungsinstitut der Diabetes Akademie Mergentheim
Organization: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Other Study IDs: NH082018_2
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2; Depressive Symptoms; Stress, Psychological; Glucose, High Blood
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — HbA1c; Cortisol; Markers of inflammation (hsCRP, IL-6, IL-1Ra, IL-18)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No DD or DS: No diabetes distress or depressive symptoms reported (CES-D < 22, PAID < 40)
- DD without DS: Diabetes distress but no depressive symptoms reported (CES-D < 22, PAID ≥ 40)
- DS without DD: Depressive symptoms but no diabetes distress reported (CES-D ≥ 22, PAID < 40)
- DD and DS: Both diabetes distress and depressive symptoms reported (CES-D ≥ 22, PAID ≥ 40)

SUMMARY:
DIA-LINK2 is a prospective observational study analysing longitudinal associations and mediating links between diabetes distress (DD), depressive symptoms (DS) and glycaemic outcomes in people with type 2 diabetes (T2DM). A total of 200 people with T2DM with different levels of DD and DS are to be enrolled.

At baseline, all participants are assessed for DD and DS, psychological and stress-related variables, self-reported self-management, HbA1c and inflammatory markers.

This is followed by a 4-week ambulatory assessment period including continuous glucose monitoring (CGM), continuous activity tracking and daily event sampling regarding sleep, stress levels, mood and diabetes-related issues; additionally, cortisol levels are assessed on four days within this period.

Three months after baseline, a follow-up assessment covers DD and DS levels, stress-related variables, self-reported self-management, HbA1c and final CGM assessment.

The analyses aim to establish risk factors/protective factors regarding DD and DS, their relative impact on glycaemic outcomes and potential mediation of the associations by behavioural (e.g. self-management, physical activity), physical (e.g. heart rate variability, inflammatory activity) and mental variables (subjective stress level) in T2DM.

DETAILED DESCRIPTION:
DIA-LINK2 is a prospective observational study analysing longitudinal associations between diabetes distress (DD), depressive symptoms (DS) and glycaemic outcomes in people with type 2 diabetes (T2DM). A variety of behavioural, physical and mental variables are assessed to analyse the mediating links between DD, DS and glycaemia.

A total of 200 people with T2DM are enrolled according to DD (PAID ≥ / < 40) and DS (CES-D ≥ / < 22) scores so that four groups (n = 50 persons each) with varying levels of DD and DS are established: 1. PAID < 40 and CES-D < 22 (no DD, no DS); 2. PAID ≥ 40 and CES-D < 22 (DD, no DS); 3. PAID < 40 and CES-D ≥ 22 (DS, no DD); 4. PAID ≥ 40 and CES-D ≥ 22 (DD and DS).

At baseline, all participants are assessed for relevant psychological and stress-related variables (daily hassles, life events, diabetes-related problems and fears, coping styles, resilience, diabetes acceptance, depression) as well as self-reported diabetes self-management using validated self-report scales and interviews; HbA1c and selected markers of inflammation (hsCRP, IL-6, IL-18, IL1Ra) are analysed from venous blood samples.

This is followed by a 4-week ambulatory assessment period including continuous glucose monitoring (CGM) (to establish time in range, glucose variability and times in hypo/hyperglycaemia), continuous activity tracking regarding general activity, movement, sleep and heart rate using a wristband as well as event sampling regarding sleep quality, stress levels, mood and diabetes-related issues four times daily using a smartphone app. Additionally, salivary cortisol levels are estimated on four consecutive days (each including a morning, afternoon and night time sample) within this period.

Three months after baseline, a follow-up assessment is performed which includes self-report measures of DD and DS, stress-related variables and diabetes self-management, HbA1c estimation from venous blood samples and final CGM assessment over 14 days.

The collected data are used to analyse risk factors/protective factors regarding DD and DS, their relative impact on glycaemic outcomes and potential mediation of the associations by behavioural (e.g. self-management, physical activity), physical (e.g. heart rate variability, inflammatory activity) and mental variables (subjective stress level) in T2DM.

The findings shall be used to develop personalised interventions for people with diabetes and comorbid mental conditions (DD and DS).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Diabetes duration at least 1 year
* Age between 18 and 70 years
* Sufficient German language skills
* Informed consent
* Smartphone available

Exclusion Criteria:

* Capacity for consent lacking
* Illness with significant impairment of cognitive functioning (e.g. dementia)
* Severe somatic illness or mental disorder which interferes with study participation or might confound the results (dialysis-dependent renal failure; heart failure, i.e. New York Heart Association (NYHA) class III or IV; cancer requiring treatment; schizophrenia/psychotic disorder; bipolar disorder; severe eating disorder F50.0/F50.2; personality disorder)
* Terminal illness
* Being bedridden

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with T2DM with different levels of diabetes distress (DD) and/or depressive symptoms (DS): Four groups of n = 50 persons each reporting 1. "no DD/no DS" vs. 2. "DD/no DS" vs. 3. "DS/no DD" vs. "DD and DS".
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 3-month follow-up
  Depressive symptoms are assessed using the 20-item Center for Epidemiologic Studies Depression Scale (CES-D), covering 20 symptoms of depression. Frequencies of the symptoms during the past week are scored on a 4-point Likert scale (from 0 - "rarely or non of the time" to 3 - "most or all of the time"). Item scores are summed to a total score ranging from 0 to 60, whereby higher values reflect higher depressive symptoms. A cut-off point at ≥ 22 points (found to have the best likelihood ratio for detecting depression within the German population) is used to establish elevated depressive symptoms in this study.
Diabetes Distress | 3-month follow-up
  Diabetes Distress is assessed as using the 20-item Problem Areas In Diabetes Scale (PAID). 20 potential problems related to living with diabetes are rated on a 5-point Likert scale (from 0 - "not a problem" to 4 - "serious problem"). Item scores are summed/transformed to a total score ranging from 0 to 100, whereby higher values reflect higher diabetes distress. A cut-off point at ≥ 40 points is commonly used to establish high diabetes distress, so too in this study.
HbA1c | 3-month follow-up
  HbA1c (estimated in %-points; mmol/mol values are calculated thereof) is used as a measure of glycaemic levels during past 3 months. It is estimated from a venous blood sample using high performance liquid chromatography (Tosho G11 analyser; meeting International Federation of Clinical Chemistry and Laboratory Medicine (IFCC) standard) in this study. Higher values indicate less optimal glycaemic control, and values above 7.5% (58 mmol/mol) are considered to indicate glycaemic levels in need of improvement.

SECONDARY OUTCOMES:
"Time in range" of glucose levels | Continuous assessment over 4 weeks from baseline
  Percentage of glucose values measured using CGM ("FreeStyle Libre 2" glucose monitoring system) during 4-week ambulatory assessment which are between 70 and 180 mg/dl (out of all measured values). Note that although the expression "time in range (TIR)" suggests a time measure, this is in fact estimated as a percentage score.
Variability of glucose levels | Continuous assessment over 4 weeks from baseline
  Estimated by the coefficient of variation (range 0 to 1) of all glucose values measured using CGM ("FreeStyle Libre 2" glucose monitoring system) during the 4-week ambulatory assessment phase.
"Time in hypoglycaemia" of glucose levels | Continuous assessment over 4 weeks from baseline
  Percentage of glucose values measured using CGM ("FreeStyle Libre 2" glucose monitoring system) during 4-week ambulatory assessment phase which are below 70 mg/dl (out of all measured values). Note that although the expression "time in hypoglycaemia" suggests a time measure, this is in fact estimated as a percentage score.
"Time in hyperglycaemia" of glucose levels | Continuous assessment over 4 weeks from baseline
  Percentage of glucose values measured using CGM ("FreeStyle Libre 2" glucose monitoring system) during 4-week ambulatory assessment phase which are over 180 mg/dl (out of all measured values). Note that although the expression "time in hyperglycaemia" suggests a time measure, this is in fact estimated as a percentage score.
Activity time | Continuous assessment over 4 weeks from baseline
  Activity time (in h/day) is measured continuously during the 4-week ambulatory assessment phase using a wearable health tracker/wristband ("Garmin vivosmart 4").
Sleep time | Continuous assessment over 4 weeks from baseline
  Sleep time (in h/day) is measured continuously during the 4-week ambulatory assessment phase using a wearable health tracker/wristband ("Garmin vivosmart 4").
Heart rate (variability) | Continuous assessment over 4 weeks from baseline
  Heart rate (in beats/minute) is measured continuously during the 4-week ambulatory assessment phase using a wearable health tracker/wristband ("Garmin vivosmart 4"). Heart rate variability is calculated thereof using the coefficient of variation.
Self-reported sleep quality | Daily assessment over 4 weeks from baseline
  Sleep quality of the past night is assessed each morning during the 4-week ambulatory assessment phase using items from the Pittsburgh Sleep Quality Index (PSQI) adapted for ecological momentary assessment (EMA). Subjective sleep quality is rated on a 10-point Likert scale (0-"very poor" to 10-"very good"). Further items request total time in bed ("How many hours did you stay in bed last night?"), sleep latency ("How many minutes did it take until you fell asleep?"), number of wake-ups ("How many times did you wake up last night?") and total time awake ("If you woke up, how many minutes did you stay awake in total?"). The following aspects are estimated thereof: sleep quality; sleep latency; sleep duration; sleep efficiency (each scored from 0 to 3; higher scores indicate more problems). The scales are summed to a total from 0 to 12; higher scores reflect lower sleep quality. Scoring of the PSQI is explained elsewhere (https://www.dgsm.de/fachinformationen_frageboegen_psqi.php).
Stress level | Daily assessment over 4 weeks from baseline
  Stress level is assessed four times daily during the 4-week ambulatory assessment phase assessed using the single item "How stressed are you feeling right now?" and a Likert scale from 0 - "not at all stressed" to 10 - "very strongly stressed" in an ecological momentary assessment (EMA) survey via smartphone.
Mood: Hedonic tone | Daily assessment over 4 weeks from baseline
  Mood is assessed twice daily during the 4-week ambulatory assessment phase using selected items from the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (UMACL) in an ecological momentary assessment (EMA) survey via smartphone. 12 of the 29 UMACL items were selected based on their significant associations with glycaemic outcomes from CGM assessment (own data set); each four of them reflect positive and negative hedonic tone and energetic and tense arousal. Responses are given on a four-point Likert scale (0 - "definitely not" / 1 - "slightly not" / 2 - "slightly" / 3 - "definitely) reflecting the presence or absence of each aspects. Item scores are summed/averaged to scale scores (from 0 to 3) reflecting hedonic tone and arousal levels; higher scores reflect higher hedonic tone and arousal levels, respectively.
Mood: Arousal | Daily assessment over 4 weeks from baseline
  Mood is assessed twice daily during the 4-week ambulatory assessment phase using selected items from the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (UMACL) in an ecological momentary assessment (EMA) survey via smartphone. 12 of the 29 UMACL items were selected based on their significant associations with glycaemic outcomes from CGM assessment (own data set); each four of them reflect positive and negative hedonic tone and energetic and tense arousal. Responses are given on a four-point Likert scale (0 - "definitely not" / 1 - "slightly not" / 2 - "slightly" / 3 - "definitely) reflecting the presence or absence of each aspects. Item scores are summed/averaged to scale scores (from 0 to 3) reflecting hedonic tone and arousal levels; higher scores reflect higher hedonic tone and arousal levels, respectively.
Diabetes-specific problems | Daily assessment over 4 weeks from baseline
  Diabetes-specific problems are assessed daily during the 4-week ambulatory assessment phase using six items adapted from the Problem Areas In Diabetes Scale and additional items in an ecological momentary assessment (EMA) survey via smartphone. Responses are given on a Likert scale from 0 - "not at all" to 10 - "very strong". Item scores are averaged to a scale ranging from 0 to 10, whereby higher scores indicate greater problems.
Cortisol | 2 weeks after baseline
  Cortisol level (in μg/dl) is estimated from saliva samples collected at fixed day times (morning; afternoon; late evening) on four consecutive days (Sat/Sun/Mon/Tue) during ambulatory assessment period. Collection date within 4 week-period is from the beginning of the third week (approx. 2 weeks after baseline). Samples are analysed using electrochemiluminescence (Cobas 6000 analyser).
Marker of inflammation #1: high sensitivity C-reactive protein (hsCRP) | Baseline
  Estimated from venous blood sample (fasting blood collection) in mg/dl.
Marker of inflammation #2: interleukin-6 (IL-6) | Baseline
  Estimated from venous blood sample (fasting blood collection) in pg/ml.
Marker of inflammation #3: interleukin-18 (IL-18) | Baseline
  Estimated from venous blood sample (fasting blood collection) in pg/ml.
Marker of inflammation #4: interleukin-1 receptor antagonist (IL-1Ra) | Baseline
  Estimated from venous blood sample (fasting blood collection) in pg/ml.

OTHER OUTCOMES:
Coping with stress | Baseline
  Coping styles regarding stressful events are assessed at baseline using the 21-item short form of the Coping Inventory for Stressful Situations (CISS-21). The scale enables estimation of three scale scores reflecting task-oriented coping, emotion-oriented coping and avoidance coping (each seven items). Responses are given on a five-point Likert scale (1 - "not at all" to 5 - "very much"). Item scores are summed to scale scores ranging from 7 to 35, whereby higher scores reflect higher use of the corresponding coping style. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Resilience | Baseline
  Resilience is assessed at baseline using the Resilience Scale (RS-13). Its 13 items are scored on a 7-point Likert scale (from 1 - "I do not agree" to 7 - "I fully agree"). Item scores are summed to a total score ranging from 13 to 91, whereby higher scores indicate greater resilience. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Life events | Baseline
  Critical life events during the past 12 months are assessed at baseline using the German "Fragebogen zu Kritischen Lebensereignissen (FKL)" (Questionnaire for Critical Life Events FKL). Emotional distress related to each of 27 possible events which occured during the past 12 months is rated on a 3-point scale (from 0 - "not at all distressing" to 2 - "very much distressing"), and scores are summed to a total score reflecting the burden of recent life events (range from 0 to 54, with higher values reflecting higher burden). Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Diabetes acceptance | Baseline
  Diabetes acceptance is assessed at baseline using a 10-item short form of the Diabetes Acceptance Scale (DAS). Each items is scored on a 3-point Likert scale from 0 - "never true for me" to 3 - "always tue for me". Items scores are summed to a total score (from 0 to 30); higher scores reflect higher diabetes acceptance. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Diabetes self-management | Baseline
  Diabetes self-management is assessed at baseline using the revised version of the Diabetes Self-Management Questionnaire (DSMQ), a 27-item scale reflecting different behaviours/activities related to the self-management of the condition during the past eight weeks. Each item is scored on a 4-point Likert scale (from 0 - "does not apply to me" to 3 - "applies to me very much"), and items scores are summed/transformed to a total score (range 0 to 10) reflecting overall diabetes self-management. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Diabetes-specific problems | Baseline
  Diabetes-specific problems are assessed at baseline using the Diabetes Distress Scale (DDS), a 17-item scale reflecting diverse problems related to living with diabetes. Items scores (from 1 - "not a problem" to 6 - "a very serious problem") are summed and averaged to a total ranging from 0 to 6 with higher values reflecting more problems. Subscale scores reflecting emotional burden, regimen-related distress, physician-related distress and interpersonal distress can also be calculated. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Fear of hypoglycaemia | Baseline
  Fear of hypoglycaemia is assessed at baseline using the 11-item short form of the Hypoglycaemia Fear Survey-II (HFS-II). The occurence of eleven hypoglycaemia-related worries and avoidance behaviours during the past four weeks is rated on a five-point Likert Scale (0 = never to 4 - "almost always"). Item scores are summed to a total score ranging from 0 to 44, whereby higher values indicate higher fear of hypoglycaemia. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).
Fear of diabetes complications | Baseline
  Fear of diabetes complications is at baseline assessed using a 6-item short form of the Fear of Complications Questionnaire (FCQ). The questionnaire requests the frequencies of worries and fears regarding risks of developing long-term complications of diabetes. Each item is rated on a four-point Likert Scale (0 = never/rarely to 3 - "very often"). Item scores are summed to a total score ranging from 0 to 18, whereby higher values indicate higher fear of diabetes complications. Note: This outcome variable is assessed to be used as a mediator or moderator or control factor in the analyses of associations between primary and secondary outcome variables (e.g. between diabetes distress and glycaemic levels).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of the Diabetes Academy Mergentheim, Diabetes Center Mergentheim, Bad Mergentheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitt A, Ehrmann D, Kuniss N, Muller N, Kulzer B, Hermanns N. Assessing fear of complications in people with type 1 and type 2 diabetes with the Fear of Diabetes Complications Questionnaire. Health Psychol. 2023 Sep;42(9):674-685. doi: 10.1037/hea0001304. Epub 2023 Jul 27. PMID 37498716